CLINICAL TRIAL: NCT07164807
Title: Comparative Efficacy of Varying Concentrations of Methylene Blue Combined With Ropivacaine for Postoperative Analgesia Following Milligan-Morgan Hemorrhoidectomy: A Single-Center, Prospective, Open-Label, Randomized, Parallel-Controlled Trial
Brief Title: Efficacy of Methylene Blue Plus Ropivacaine for Post-Hemorrhoidectomy Pain.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Affiliated Hospital of Putian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHPuTianU-011
Record Dates: First submitted 2025-08-29; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Mixed Hemorrhoids; Milligan-Morgan Hemorrhoidectomy; Methylene Blue
MeSH Terms: interventions — Methylene Blue; Ropivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Concentration Methylene Blue with Ropivacaine Group (Experimental): Intervention: Perianal subcutaneous injection of 0.1% methylene blue solution (Formulation: 0.5 mL of 1% methylene blue with 4.5 mL ropivacaine hydrochloride injection).
  Interventions: Drug: Methylene Blue (0.3%) with Ropivacaine Hydrochloride (0.75%)
- Low-Concentration Methylene Blue with Ropivacaine (Experimental): Intervention: Perianal subcutaneous injection of 0.3% methylene blue solution (Formulation: 1.5 mL of 1% methylene blue with 3.5 mL ropivacaine hydrochloride injection).
  Interventions: Drug: Methylene Blue (0.1%) with Ropivacaine Hydrochloride (0.75%)
- Ropivacaine hydrochloride injection Group (No Intervention): Postoperative protocol: No routine preemptive analgesia administered.

INTERVENTIONS:
Drug: Methylene Blue (0.3%) with Ropivacaine Hydrochloride (0.75%) — Perianal subcutaneous injection of 0.3% methylene blue solution (Formulation: 1.5 mL of 1% methylene blue with 3.5 mL ropivacaine hydrochloride injection).
  Arms: High-Concentration Methylene Blue with Ropivacaine Group
Drug: Methylene Blue (0.1%) with Ropivacaine Hydrochloride (0.75%) — Perianal subcutaneous injection of 0.1% methylene blue solution (Formulation: 0.5 mL of 1% methylene blue with 4.5 mL ropivacaine hydrochloride injection).
  Arms: Low-Concentration Methylene Blue with Ropivacaine

SUMMARY:
Revised Translation (Academic English):

As one of the most prevalent anorectal disorders, mixed hemorrhoids continue to rely on the Milligan-Morgan hemorrhoidectomy as the gold-standard surgical approach. While this technique demonstrates well-established efficacy, managing acute postoperative pain-particularly during the critical 24-72-hour peak pain window-remains a persistent clinical challenge. Recent advancements in multimodal analgesia have highlighted the potential of local nerve blockers, with methylene blue (MB) gaining scientific interest due to its prolonged analgesic properties. This randomized controlled study systematically evaluates the synergistic analgesic effects of gradient concentrations of MB combined with ropivacaine (ROP) following Milligan-Morgan procedures. Therapeutic safety profiles were validated through dual-dimensional monitoring of Visual Analog Scale (VAS) scores and complication rates, aiming to establish evidence-based optimal dosing protocols and refine perioperative pain management strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years.
2. Diagnosed with Grade III-IV hemorrhoids according to the Goligher classification.
3. Scheduled to undergo standard Milligan-Morgan hemorrhoidectomy.
4. Procedure performed under spinal anesthesia alone.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Current immunotherapy or coagulopathies.
3. Contraindications to any protocol-specified agents (e.g., history of severe allergic reactions to methylene blue or ropivacaine).
4. Concurrent anorectal pathologies (e.g., perianal abscess, anal fistula, fecal incontinence).
5. Comorbid systemic conditions (e.g., cardiac/hepatic/renal insufficiency, diabetes mellitus, coagulopathy, peptic ulcer disease).
6. Incomplete perioperative documentation.
7. Inability to comply with follow-up protocols.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Numerical Rating Scale (NRS) Pain Scores | Within 30 days after surgery
  Assessment timepoints: At postoperative days 1, 2, 3, 4, 5days, 2 weeks, and 1 month.0 usually means "no pain."10 means "the worst pain imaginable.
Total Postoperative Analgesic Consumption | Within 30 days after surgery
  Metric: Cumulative dosage of rescue analgesics (e.g., NSAIDs or opioids) administered during the follow-up period.
Postoperative Quality of Life (QoL) Metrics | Within 30 days after surgery
  Postoperative QoL metrics are standardized tools (questionnaires, surveys) used to measure a patient's overall well-being and functional status after a surgical procedure.patients rate their overall health from 0 (worst) to 100 (best).

SECONDARY OUTCOMES:
Incidence of Postoperative Complications | Within 30 days after surgery
  Documented adverse events:urinary retention,secondary hemorrhage,perianal edema,secondary infection,pruritus and other procedure-related morbidities.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Putian University, Putian, China